CLINICAL TRIAL: NCT02902289
Title: Bioequivalence Study of a New Formulation of Ibuprofen 200 mg/5 mL Oral Suspension vs. the Reference Product MOMENT 200 mg Coated Tablet in Healthy Volunteers
Brief Title: Bioequivalence Study of Ibuprofen 200 mg/5 mL Oral Suspension vs. MOMENT 200 mg Coated Tablet
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Aziende Chimiche Riunite Angelini Francesco S.p.A (Industry)
Collaborators: Cross Research S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 070(Q)HO15411; CRO-PK-15-306 (Other: CROSS Research S.A., Phase I Unit)
Record Dates: First submitted 2016-09-07; First posted 2016-09-15 (Estimated); Last update posted 2016-09-15 (Estimated); Status verified 2016-07

CONDITIONS: Healthy
Keywords: Bioequivalence; Ibuprofen 200 mg/5 ml; Moment 200 mg coated tablet; Oral Suspension
MeSH Terms: interventions — Ibuprofen; Suspensions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ibuprofen 200 mg/5 mL oral suspension (Experimental): Single dose of 1 ibuprofen 200 mg/5 mL stick administered under fasting conditions in two consecutive periods, with a wash-out interval of at least 7 days between consecutive administrations.
  Interventions: Drug: Ibuprofen 200 mg/5 mL oral suspension
- MOMENT 200 mg coated tablet (Active Comparator): Single dose of 1 MOMENT 200 mg coated tablet administered under fasting conditions in two consecutive periods, with a wash-out interval of at least 7 days between consecutive administrations.
  Interventions: Drug: MOMENT 200 mg coated tablet

INTERVENTIONS:
Drug: Ibuprofen 200 mg/5 mL oral suspension
  Arms: Ibuprofen 200 mg/5 mL oral suspension
Drug: MOMENT 200 mg coated tablet
  Arms: MOMENT 200 mg coated tablet

SUMMARY:
The main objective of the study is to evaluate the bioequivalence of a new formulation of ibuprofen 200 mg/5 mL oral suspension vs. the marketed reference product MOMENT 200 mg coated tablet, when administered under fasting conditions as single oral dose to healthy male and female volunteers, in two consecutive study periods.

ELIGIBILITY:
Inclusion Criteria:

To be enrolled in this study, subjects must fulfil all these criteria:

1. Informed consent: signed written informed consent before inclusion in the study
2. Sex and Age: males/females, 18-55 years old inclusive
3. Body mass index (BMI): 18.5-30 kg/m2 inclusive
4. Vital signs: systolic blood pressure (SBP) 100-139 mmHg, diastolic blood pressure (DBP) 50-89 mmHg, heart rate (HR) 50-90 bpm, measured after 5 min at rest in the sitting position
5. Full comprehension: ability to comprehend the full nature and purpose of the study, including possible risks and side effects; ability to co-operate with the investigator and to comply with the requirements of the entire study
6. Contraception and fertility (females only): females of child-bearing potential must be using at least one of the following reliable methods of contraception:

   1. Hormonal oral, implantable, transdermal, or injectable contraceptives for at least 2 months before the screening visit
   2. A non-hormonal intrauterine device [IUD] or female condom with spermicide or contraceptive sponge with spermicide or diaphragm with spermicide or cervical cap with spermicide for at least 2 months before the screening visit
   3. A male sexual partner who agrees to use a male condom with spermicide
   4. A sterile sexual partner Female participants of non-child-bearing potential or in post-menopausal status for at least 1 year will be admitted. For all female subjects, pregnancy test result must be negative at screening and day -1.

Exclusion Criteria:

1. Electrocardiogram (12-leads, supine position): clinically significant abnormalities
2. Physical findings: clinically significant abnormal physical findings which could interfere with the objectives of the study
3. Laboratory analyses: clinically significant abnormal laboratory values indicative of physical illness
4. Allergy: ascertained or presumptive hypersensitivity to the active principle and/or formulations' ingredients or related drugs, namely non-steroidal anti-inflammatory agents (NSAIDs); history of anaphylaxis to drugs or allergic reactions in general, which the investigator considers may affect the outcome of the study
5. Diseases: history of significant renal, hepatic, gastrointestinal (in particular gastroduodenal ulcer and bleeding), cardiovascular, respiratory (in particular asthma), skin, haematological, endocrine or neurological diseases that may interfere with the aim of the study
6. Medications: medications, including over the counter (OTC) (in particular ibuprofen) medications and herbal products for 2 weeks before the start of the study. Hormonal contraceptives for females will be allowed
7. Investigative drug studies: participation in the evaluation of any investigational product for 3 months before this study. The 3-month interval is calculated as the time between the first calendar day of the month that follows the last visit of the previous study and the first day of the present study
8. Blood donation: blood donations for 3 months before this study
9. Drug, alcohol, caffeine, tobacco: history of drug, alcohol [>1 drink/day for females and >2 drinks/day for males, defined according to USDA Dietary Guidelines 2015-2020 (10)], caffeine (>5 cups coffee/tea/day) or tobacco abuse (≥10 cigarettes/day)
10. Drug test: positive result at the drug test at screening or day-1
11. Alcohol test: positive alcohol breath test at day -1
12. Diet: abnormal diets (<1600 or >3500 kcal/day) or substantial changes in eating habits in the 4 weeks before this study; vegetarians
13. Pregnancy (females only): positive or missing pregnancy test at screening or day -1,pregnant or lactating women

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2016-06; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Cmax of (S)-ibuprofen after single dose administration under fasting conditions of test and reference formulations containing racemic ibuprofen. | 0 (pre-dose), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10 hours post-dose
  Maximum plasma concentration (μg/ml)
AUC(0-t) of (S)-ibuprofen after single dose administration under fasting conditions of test and reference formulations containing racemic ibuprofen. | 0 (pre-dose), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10 hours post-dose
  Area under the plasma concentration-time curve from administration time to the time (t) of the last measurable concentration (Ct ), calculated with the linear trapezoidal method (μg*h/ml)

SECONDARY OUTCOMES:
Peak drug concentration (Cmax) of racemic ibuprofen and (R)-ibuprofen after single dose administration under fasting conditions of test and reference formulations | 0 (pre-dose), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10 hours post-dose
Area under the concentration-time curve from time zero to time t (AUC(0-t)) of racemic ibuprofen and (R)-ibuprofen after single dose administration under fasting conditions of test and reference formulations | 0 (pre-dose), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10 hours post-dose
Area under the concentration-time curve from time zero to time t (AUC(0-t)) ratio of the two enantiomers (S/R) after single dose administration under fasting conditions of test and reference formulations | 0 (pre-dose), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10 hours post-dose
  Area under the concentration-time curve extrapolated to infinity, calculated, if feasible, as AUC(0-t) + Ct/λz, where Ct is the last measurable drug concentration (μg*h/ml)
Area under the concentration vs. time curve up to infinity (AUC(0-∞)) of ibuprofen racemate and of (S)-ibuprofen and (R)-ibuprofen after single dose administration under fasting conditions of test and reference formulations | 0 (pre-dose), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10 hours post-dose
Extrapolated area calculated as (AUC(0-∞) - AUC(0-t))/AUC(0-∞) (residual area) of ibuprofen racemate and of (S)-ibuprofen and (R)-ibuprofen after single dose administration under fasting conditions of test and reference formulations | 0 (pre-dose), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10 hours post-dose
Time to achieve Cmax (Tmax) of ibuprofen racemate and of (S)-ibuprofen and (R)-ibuprofen after single dose administration under fasting conditions of test and reference formulations | 0 (pre-dose), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10 hours post-dose
Half-life lambda z (/t1/2,z) of ibuprofen racemate and of (S)-ibuprofen and (R)-ibuprofen after single dose administration under fasting conditions of test and reference formulations | 0 (pre-dose), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10 hours post-dose
Apparent First order terminal rate constant (λz) of ibuprofen racemate and of (S)-ibuprofen and (R)-ibuprofen after single dose administration under fasting conditions of test and reference formulations | 0 (pre-dose), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10 hours post-dose
Time Until First Nonzero Concentration (tlag) of ibuprofen racemate and of (S)-ibuprofen and (R)-ibuprofen after single dose administration under fasting conditions of test and reference formulations | 0 (pre-dose), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10 hours post-dose
Treatment-Emergent Adverse Event (TEAEs), vital signs (BP, HR), physical examination, body weight and laboratory parameters | 0 (pre-dose), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10 hours post-dose
A descriptive evaluation of palatability for the test formulation will be performed. Smell, taste and texture parameters will be evaluated immediately after drug administration through a 5-point rating scale. | 0 (pre-dose), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Milko Radicioni, MD, Principal Investigator — Cross Research S.A.
Locations (1):
- CROSS Research S.A., Phase I Unit, Arzo, Switzerland, Switzerland

IPD SHARING:
Plan to Share IPD: No